CLINICAL TRIAL: NCT06722651
Title: Randomized Controlled Clinical Study to Evaluate the Novel Netrod™ Renal Denervation System and the Impact of Sham vs Open-Label Control in European Patients With Uncontrolled Primary Hypertension in the Absence of Hypertensive Medication
Brief Title: EuroNetrod HTN OFF-Med Study of Renal Denervation With NetrodTM Six-electrode Radiofrequency RDN System
Acronym: EuroNetrod
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This decision aims to concentrate resources on accelerating the development of the next generation of the NetrodTM RDN System.This reflects a broader strategy to advancing more effective solutions for physicians and patients.
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGL-01
Record Dates: First submitted 2024-11-15; First posted 2024-12-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Uncontrolled Hypertension
Keywords: Renal denervation (RDN); Radiofrequency renal denervation; Sympathetic nervous system; Interventional therapy; Interventional cardiology; Device-based therapy; Renal artery denervation; Blood pressure; Resistant Hypertension; Refractory Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the RDN procedure, sham procedure, or open-label control (where patients do not receive any procedure and are off medication until primary endpoint measurement). After primary endpoint measurements at Month 3, patients in the sham and open-label control groups will have the option to receive the RDN procedure, referred to as "crossover patients."
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Renal Denervation (Experimental): Renal angiogram and Renal Denervation procedure
  Interventions: Device: Netrod™ six-electrode radiofrequency renal denervation system
- Sham Control group (Sham Comparator): Renal angiogram followed by Sham procedure
  Interventions: Device: Sham Procedure
- Open-label Control group (No Intervention): The patient will not undergo either the renal angiogram or the RDN procedure.

INTERVENTIONS:
Device: Netrod™ six-electrode radiofrequency renal denervation system — Netrod™ renal denervation (RDN) system, which is indicated for the treatment of uncontrolled hypertension. It consists of the following two components:
  * Netrod™ Six-Electrode Basket Radiofrequency Renal Denervation Catheter and
  * Netrod™ Renal Denervation Radiofrequency Generator The catheter's electrodes deploy into a self-adaptive basket structure, optimizing contact with the vessel wall for effective ablation.
  Arms: Renal Denervation
Device: Sham Procedure — Patients will be remained on the catheterization table for at least 20 min prior to sheath removal.
  Arms: Sham Control group

SUMMARY:
This randomized controlled investigation aims to evaluate the efficacy and safety of the Netrod™ RDN system in patients with uncontrolled primary hypertension in the absence of antihypertensive medication, comparing the outcomes between renal denervation, sham procedure, and open-label control groups.

DETAILED DESCRIPTION:
This is a prospective, multi-center, blinded, three-arm randomized controlled study to demonstrate the effectiveness and safety of the Netrod™ RDN system for treating treating patients with uncontrolled primary hypertension in the absence of antihypertensive medications. This clinical investigation will enroll 260 patients in Europe. Patients with uncontrolled primary hypertension (office BP ≥150/90 mmHg and <180/110 mmHg) who are willing to discontinue antihypertensive medications will be screened after providing informed consent.

All eligible patients will undergo a medication washout period of at least three weeks, and those who continue to meet the eligibility requirements will be randomized in a 2:1:1 ratio to one of three groups: renal denervation (RDN), a sham procedure (renal artery angiogram only), or an open-label group (not undergoing the renal angiogram).

All subjects randomized to either the treatment or sham procedure groups will be evaluated at hospital discharge. All subjects will be evaluated at 1 and 3 months post-procedure. Additionally, patients who undergo the RDN procedure will also be evaluated at 12, 24, and 36 months post-procedure. All subjects will remain off antihypertensive medications until the primary endpoint is assessed at the 3-month follow-up visit, after which antihypertensive medications may be reintroduced.

Patients in the RDN and sham-control groups, as well as all clinical follow-up assessors, will be blinded to the treatment allocation. The primary efficacy endpoint is the change in daytime ambulatory systolic blood pressure (ASBP) from baseline at three months post-procedure. The primary safety endpoint is the periprocedural major adverse event (MAE) rate at 30 days post-procedure.

Subjects enrolled in the sham and open-label control groups may cross over to RDN at three months. Those who cross over will restart the follow-up schedule post-RDN procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age ≥18 years or minimum age as required by local regulations and ≤80 years old at time of consent
2. Subject with hypertension who has an office BP of ≥150/90 mmHg and <180/110 mmHg (meet both SBP and DBP criteria) at screening V3 and mean daytime ASBP ≥140 mmHg and <170 mmHg by 24-hour ABPM at Screening V3
3. Subject or his/her legal representative must sign an IEC/REB-approved ICF for the study
4. Subject is willing to discontinue current antihypertensive medications at Screening V1 through the 3-month follow-up visit

Exclusion Criteria:

1. 1. Subject who is pregnant, nursing or planning to become pregnant during the course of the study
2. Subject with unilateral or bilateral renal artery that are not suitable for ablation procedure (renal artery stenosis more than 50%, renal aneurysm, renal artery abnormality, renal artery diameter <3 mm or treatable segment length <20 mm)
3. Subject with single-kidney or history of kidney transplant
4. Subject with history of renal artery intervention (PTA or stenting) or RDN
5. Subject with any conditions that may affect the accuracy of blood pressure measurement: such as the diameter of the upper arm is too large for the cuff, or arrhythmia, etc.
6. Subject with known secondary hypertension
7. Subject with eGFR <40 mL/min/l.73m²
8. Subject with history of hospitalization for hypertensive emergency within past year
9. Subject with type I diabetes mellitus
10. Subject with primary pulmonary hypertension
11. Subject with history of bleeding diathesis and haematological disorders or coagulopathy
12. Subject with recent history of any embolism within 6 months
13. Subject with history of coronary artery intervention, unstable angina or myocardial infarction
14. Subject with stable angina and therefore treated anti-anginal medication (betablockers, calcium antagonists, long-acting nitrates)
15. Subject with history of abdominal aortic aneurysm
16. Subject with atrial fibrillation or history of atrial fibrillation in the last 3 years or on rhythm control medication for arrhythmia
17. Subject with a history of ventricular fibrillation or ventricular tachycardia
18. Subject known with serum HIV-positive
19. Subject who is allergic to contrast agents and not responding to preventive medication
20. Subject with acute or severe systemic infections
21. Subject with mental illness or any psychological problems that may interfere with participating in the study
22. Subject with history of stroke or transient ischemic attack (TIA)
23. Subject with malignant tumors or end-stage disease
24. Subject with severe PAD along the access path to renal arteries, including abdominal aneurysm
25. Subject with severe heart valve stenosis or regurgitation
26. Subject with heart failure requiring medications (i.e. ACE/ARB, SGTL2i, diuretics).
27. Subject with uncontrolled hyperthyroidism or hypothyroidism
28. Subject with severe electrolyte abnormalities, defined as values above and below the limits of normal (ULN) on repeated measurements despite normalization efforts, or with liver function abnormalities, defined as 2 > ULN
29. Subject who requires mechanical ventilation other than CPAP for sleep apnea
30. Subject with a implanted pacemaker or ICD/CRT device
31. Subject with a history of major surgery or trauma within 30 days prior to enrolment
32. Subject who has planned surgery or cardiovascular intervention within the next 12 months
33. Subject who is participating in other drug or medical device clinical investigations
34. Subject who has known drug or alcohol dependence, difficulty to understand the clinical investigation protocol, inability/unwillingness to follow the clinical investigation protocol
35. Subject who is unsuitable to participate in this study in the opinion of investigators
36. Subjects who are incapacitated or unable to provide informed consent due to cognitive impairment, mental illness, or other conditions that affect their decision-making capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Mean daytime ambulatory systolic blood pressure | From baseline at Screening Visit 2 to Month 3 post-procedure
  Between-group difference in baseline adjusted change in mean daytime ambulatory systolic blood pressure (ASBP) at 3 months compared to baseline measured by 24 hours ambulatory blood pressure monitoring (ABPM) (RDN vs sham vs open-label).
Periprocedural major adverse event (MAE) rate | At 30 days post-procedure
  Periprocedural major adverse event (MAE) rate, defined as a composite of the following events at 30 days post procedure:
  * All-cause mortality
  * End-stage renal disease (ESRD) defined as stage 5 CKD (eGFR < 15 mL/min/l.73m²) or hemodialysis
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation or dissection requiring intervention
  * Major vascular complications requiring medical or surgical intervention
  * Hospitalization for hypertensive crisis (unless clearly demonstrated to be associated with non-adherence with antihypertensive medications in the subjects on escape medication)
  * New renal artery stenosis > 70% (must be confirmed by angiography)

SECONDARY OUTCOMES:
Office blood pressure (BP) and home BP | From baseline at Screening Visit 2 to Month 1, 3, 12, 24 and 36 post-procedure
  Changes from baseline in office blood pressure (BP) and home BP at 1- and 3-month post procedure for all enrolled subjects, and 12-, 24- and 36-month post procedure for the subjects who underwent RDN
Mean ambulatory BP including 24-hour ASBP and ADBP, daytime and nighttime SBP and DBP | From baseline at Screening Visit 2 to Month 1, 3, 12, 24 and 36 post-procedure
  Changes from baseline in mean ambulatory BP including 24-hour ASBP and ADBP, daytime and nighttime SBP and DBP measured by 24-hour ABPM at 1-, 3-month for all enrolled subjects, and 12-, 24- and 36-month for the subjects who underwent RDN.
Percentage of patients with office systolic BP (SBP) within the target range (SBP <140 mmHg) | At Month 3, 12, 24 and 36 post-procedure
  Percentage of patients with office systolic BP (SBP) within the target range (SBP <140 mmHg) at 3-month post procedure for all enrolled subjects, and 12-, 24- and 36-month post procedure for the subjects who underwent RDN
Percentage of patients with office systolic blood pressure (SBP) within the target range (SBP <130 mmHg) | At Month 3, 12, 24 and 36 post-procedure
  Percentage of patients with office systolic blood pressure (SBP) within the target range (SBP <130 mmHg) at 3-month post procedure for all enrolled subjects, and 12-, 24- and 36-month post procedure for the subjects who underwent RDN
Percentage of patients with mean ambulatory systolic blood pressure (ASBP) within the target range (SBP <130 mmHg) | At Month 3, 12, 24 and 36 post-procedure
  Percentage of patients with mean ambulatory systolic blood pressure (ASBP) within the target range (SBP <130 mmHg) at 3-month post procedure for all enrolled subjects, and 12-, 24- and 36-month post procedure for the subjects who underwent RDN
The proportion of ambulatory SBP decreased by 5 and 10 mmHg | At Month 3 post-procedure
  The proportion of ambulatory SBP decreased by 5 and 10 mmHg at 3-month post procedure
Safety event rates | At Month 3 post-procedure
  The following safety event rates to 3-month post procedure for all enrolled subjects, and the following event rates at 12-, 24- and 36-month post procedure for the subjects who underwent RDN procedure:
  * All-cause mortality
  * End-stage renal disease (ESRD) defined as stage 5 CKD (eGFR < 15 mL/min/l.73m²)
  * ≥50% decline in eGFR or >50% increase in serum creatinine from baseline
  * New myocardial infarction or acute coronary syndrome (ACS)
  * New stroke or CVA
  * Renal artery reintervention
  * New renal artery stenosis > 70% confirmed by angiography
  * Hospitalization for hypertensive crisis not related to confirmed non-adherence of antihypertensive medications
  * Hospitalization for major cardiovascular- or hemodynamic-related events (such as heart failure or atrial fibrillation)
Device deficiency rates | At Visit 4, day 0 (procedure)
  Device deficiency rates
Quality of life changes | From baseline at Screening Visit 2 to Month 3, 12, 24 and 36 post-procedure
  Quality of life changes at 12 months and annually through 3 years post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, Prof. Dr., Principal Investigator — Department of Cardiology, University Hospital Basel; Andrew Sharp, Prof., Principal Investigator — The Mater Misericordiae University Hospital
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Gao F, Ren C, Ma G, Bu P, Fu G, Chen H, Han Z, Li Y, Li J, Ma X, Hao L, Chen Y, Chen M, Chen X, Liu X, Jiang J, Yu J, Li N, Ma X, Yang B, Cong H, Wang X, Fan Q, Lv S, Wu D, Dai Q, Qiu F, Cai H, Zhou YJ. The Netrod six-electrode radiofrequency renal denervation system for uncontrolled hypertension: a sham-controlled trial. Eur Heart J. 2024 Nov 21;45(44):4761-4764. doi: 10.1093/eurheartj/ehae703. No abstract available. PMID 39431289